CLINICAL TRIAL: NCT03540381
Title: Relation Among Cholesterol Uptake Capacity Which Measure HDL Functionality, Neoatherosclerosis and Target Lesion Revascularization After Stent Implantation
Brief Title: Relation Among HDL Functionality, Neoatherosclerosis and Target Lesion Revascularization
Status: Completed | Type: Observational
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Division of Cardiovascular Medicine, Department of Internal Medicine, Assistant Professor, Kobe University
Other Study IDs: KobeU-152M816M
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease Progression
Keywords: Neoatherosclerosis; Cholesterol Uptake Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Identified neoatherosclerosis group: From the patients treated with coronary stents, the investigators functionally evaluated their HDL by measuring the CUC. the investigators also performed follow-up OCT to evaluate the presence of neoatherosclerosis. Consecutive patients were divided into two groups. The patients with neoatherosclerosis were identified neoatherosclerosis group and the remaining were not-identified neoatherosclerosis group. After that, clinical follow-up was performed to assess TLR and the investigators examined the relation between CUC, neoatherosclerosis and TLR.
  Interventions: Other: neoatherosclerosis
- Not-identified neoatherosclerosis group

INTERVENTIONS:
Other: neoatherosclerosis
  Groups: Identified neoatherosclerosis group

SUMMARY:
The aim of this study is to evaluate the relation among cholesterol uptake capacity which measure HDL functionality, neoathrosclerosis and target-lesion revascularization.

DETAILED DESCRIPTION:
Intracoronary stent implantation has markedly reduced the incidence of restenosis in patients with coronary artery disease. However, in-stent restenosis requiring target-lesion revascularization (TLR) occurs even with the use of drug-eluting stents. Emerging evidence suggests that among various potential risk factors, atherogenic progression within the neointima, "neoatherosclerosis" is one of the major contributors to TLR, and that patients' lipid profile is one of the key risk factors for the development of neoatherosclerosis.

Conversely, recent animal and human studies have demonstrated the importance of high-density lipoprotein (HDL) functionality, rather than of HDL-cholesterol levels, in the development of de novo coronary artery disease. Cholesterol efflux capacity, a measure of the ability of HDL to promote cholesterol removal from lipid-laden macrophages, was found to be inversely correlated with the incidence of cardiovascular events and was shown to improve cardiovascular risk prediction beyond that with the use of traditional coronary risk factors. Therefore, the investigators hypothesized that the HDL function of promoting cholesterol removal from lipid-laden macrophages could be associated with TLR through its effect on the process of neoatherosclerosis progression within stents.

Recently, the investigators developed a rapid cell-free assay system to directly evaluate the capacity of HDL to accept additional cholesterol; the measurement of this cholesterol uptake capacity (CUC) enables HDL functionality to be readily evaluated in our daily practice. Thus, the investigators performed this study in order to clarify the potential relationship among CUC, neoatherosclerosis, and TLR by using the novel cell-free assay system, CUC measurement, and optical coherence tomography (OCT) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary artery disease
* Patients who had undergone percutaneous coronary intervention
* Patients who had been treated with bare-metal stents, drug-eluting stents
* Patients who had successfully undergone follow-up OCT for the target stents >6 months after stenting.

Exclusion Criteria:

* The stent was implanted in the left main trunk
* OCT images were of insufficient quality

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consist of the consecutive patients who have undergone coronary-artery OCT. the investigators performed OCT for these reasons: (1) planned follow-up coronary angiography and OCT as routine stent follow-up or due to other study protocols, regardless of symptoms; (2) evidence of myocardial ischemia, such as silent myocardial ischemia, stable angina, or acute coronary syndrome; or (3) planned follow-up angiography for other stent segments. Exclusion criteria for OCT were (1) anatomically unsuitable target artery for OCT, according to previously described criteria; (2) apparent congestive heart failure; (3) renal insufficiency with baseline creatinine level of ≥2.0 mg/dL except for under hemodialysis; or (4) no written informed consent from the patient.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Cholesterol Uptake Capacity (CUC) | an average of a year and a half
  CUC is a new rapid cell-free assay system to evaluate the functional capacity of HDL to accept additional cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Hiromasa Otake, PhD, Study Chair — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Undecided